CLINICAL TRIAL: NCT07013305
Title: Pre- and Post-Treatment Investigation of B12 and Folic Acid (Folate) Levels in Patients Receiving Antiepileptic (Anticonvulsant) Treatment for Fibromyalgia: Retrospective Study
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 03
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia (FM); Vitamin B 12 Deficiency; Folic Acid Deficiency
Keywords: Antiepileptic (anticonvulsant) drugs; Vitamin D deficiency
MeSH Terms: conditions — Fibromyalgia; Vitamin B 12 Deficiency; Folic Acid Deficiency; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibromyalgia is a rheumatological disorder characterised by chronic widespread body pain, second most common after osteoarthritis. The overall prevalence is 2-8% and it is more common in women. Diffuse body pain, fatigue, sleep and cognitive dysfunction occur. The etiology of fibromyalgia is multifactorial and occurs due to central and peripheral pain mechanisms that occur with neuroendocrine imbalance due to psychological and physical stress in people with genetic predisposition. The diagnostic criteria for fibromyalgia were updated by the American College of Rheumatology in 2016 to include a widespread body pain scale and a symptom severity scale.

Fibromyalgia treatment consists of drug (antidepressants and antiepileptics) and non-drug treatments. Pregabalin is also used in the treatment of epilepsy by blocking and modulating the α2 δ subunit of voltage-dependent calcium channels. There are studies showing that antiepileptics cause folate and vitamin B12 deficiency in epilepsy patients. In our study, we aimed to retrospectively investigate vitamin B12 and folic acid levels before and after treatment in patients with fibromyalgia using antiepileptics (anticonvulsants).

DETAILED DESCRIPTION:
After the acceptance of the study (after obtaining ethics committee approval), patients who have been followed up for at least 6 months in the physical medicine and rehabilitation outpatient clinic with a diagnosis of fibromyalgia and who use pregabalin will be evaluated retrospectively (1-year records). Blood vitamin B12 and folate (folic acid) levels of the patients before and after antiepileptics (anticonvulsants). use will be determined. Patients will be evaluated whether there is a change in vitamin B12 and folic acid levels due to antiepileptics (anticonvulsants) drug use.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years who have been diagnosed with fibromyalgia, whose vitamin B12 and folic acid levels have been analysed, who do not receive vitamin B12 and folic acid treatment, and who do not have diabetes mellitus, liver and kidney failure

Exclusion Criteria:

* Patients receiving vitamin B12 and folic acid therapy at the time of antiepileptic (anticonvulsant) drugs initiation, patients with hepatic and renal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were followed up for 6 months in the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia and who used antiepileptic (anticonvulsant) drugs will be retrospectively evaluated for the 6 months period (June-December 2024) before the ethics committee approval was obtained. Blood vitamin B12 and folate (folic acid) levels of the patients before and after antiepileptic drug use will be determined. Patients will be evaluated whether there is a change in vitamin B12 and folic acid levels depending on drug use.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 level analysed before treatment (pre-treatment) (retrospective) | Within 1 month
  Vitamin B12 level (pg/mL) among the laboratory parameters analysed before antiepileptic treatment (pre-treatment) for fibromyalgia will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
Vitamin B12 level analysed after treatment (post-treatment) (retrospective) | Within 1 month
  Vitamin B12 level (pg/mL) among the laboratory parameters analysed after antiepileptic treatment (post-treatment) for fibromyalgia will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
Folic acid level analysed before treatment (pre-treatment) (retrospective) | Within 1 month
  Folic acid level (ng/mL), one of the laboratory parameters analysed before antiepileptic treatment for fibromyalgia (pre-treatment), will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
Folic acid level analysed after treatment (post-treatment) (retrospective) | Within 1 month
  Folic acid level (ng/mL), one of the laboratory parameters analysed after antiepileptic treatment for fibromyalgia (post-treatment), will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.

SECONDARY OUTCOMES:
25-OH Vitamin D level analysed before treatment (pre-treatment) (retrospective) | Within 1 month
  D vitamini (25-OH Vitamin D) (ng/mL) among the laboratory parameters analysed before antiepileptic treatment (pre-treatment) for fibromyalgia will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.
25-OH Vitamin D level analysed after treatment (post-treatment) (retrospective) | Within 1 month
  25-OH Vitamin D (ng/mL) among the laboratory parameters analysed after antiepileptic treatment (post-treatment) for fibromyalgia will be screened retrospectively. Patients who applied to the physical medicine and rehabilitation clinic with a diagnosis of fibromyalgia in the last 6 months (June-December 2024) before the ethics committee application date, who were followed up with this diagnosis and started antiepileptic treatment will be screened within 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

REFERENCES:
- [Background] Mula M, Sander JW. Negative effects of antiepileptic drugs on mood in patients with epilepsy. Drug Saf. 2007;30(7):555-67. doi: 10.2165/00002018-200730070-00001. PMID 17604407
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Talotta R, Bazzichi L, Di Franco M, Casale R, Batticciotto A, Gerardi MC, Sarzi-Puttini P. One year in review 2017: fibromyalgia. Clin Exp Rheumatol. 2017 May-Jun;35 Suppl 105(3):6-12. Epub 2017 Jun 28. PMID 28681712
- [Result] Aslan K, Bozdemir H, Unsal C, Guvenc B. The effect of antiepileptic drugs on vitamin B12 metabolism. Int J Lab Hematol. 2008 Feb;30(1):26-35. doi: 10.1111/j.1751-553X.2007.00910.x. PMID 18190464
- [Result] Linnebank M, Moskau S, Semmler A, Widman G, Stoffel-Wagner B, Weller M, Elger CE. Antiepileptic drugs interact with folate and vitamin B12 serum levels. Ann Neurol. 2011 Feb;69(2):352-9. doi: 10.1002/ana.22229. Epub 2011 Jan 19. PMID 21246600